CLINICAL TRIAL: NCT03713801
Title: Metformin and Vaccine Response in Older Adults
Brief Title: Impact of Metformin on Immunity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20180171H
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Aging; Vaccine Response Impaired
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Dosage is increased over the first 3 weeks up to three 500 mg tablets a day at 3 weeks, then continued on 3 tablets daily for a further 9 weeks.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo tablet dosage is increased over the first 3 weeks up to three tablets a day at 3 weeks, then continued on 3 tablets daily for a further 9 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Total daily dose titrated up to 1500 mg po q day over the course of 3 weeks and continued for a total exposure of 12 weeks.
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo — Placebo tablets titrated up to 3 tablets over the course of 3 weeks and then continued as 3 daily for a total exposure of 12 weeks
  Other Names: Placebo oral tablet
  Arms: Placebo

SUMMARY:
To determine whether metformin (MET) can improve the immune response to the pneumococcal conjugate vaccine (PCV-13) in older adults.

DETAILED DESCRIPTION:
The objective of this study is to determine whether metformin (MET) can improve the immune response to the pneumococcal conjugate vaccine (PCV-13) in older adults, and if this effect is mediated by the gut microbiota.

The proposed research projects will provide the necessary pilot data for future, more definitive, studies that will evaluate the impact of immunomodulatory therapies, such as MET therapy, on the aging immune system. The specific aims are:

Aim 1. Compare PCV13 vaccine response in elderly adults (≥63 years of age) treated with MET vs. placebo. For this study, 50 elderly volunteers will be enrolled and randomly assigned to receive MET or placebo. The hypothesis that MET can improve vaccine responsiveness by measuring serotype-specific IgG concentrations before and 30 days after PCV13 administration will be tested.

Aim 2. Determine whether the frequencies of immunophenotypes differ between elderly adults treated with MET vs. placebo. The mechanisms of MET's effect on the immune system by comparing immunophenotypes of MET and placebo groups between baseline and prior to PCV13 and between baseline and 30 days after PCV13 administration will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age 63 to 89 years of age
2. No history of pneumococcal vaccinations
3. Able to take oral medications
4. Able to provide informed consent
5. Not currently taking metformin

Exclusion Criteria:

1. Previous vaccination with any pneumococcal vaccine
2. Metformin within the last 6 months
3. Contraindication for PCV13
4. History of severe adverse reaction associated with any vaccine component
5. Residence in long-term care facility
6. Diagnosis of diabetes (diagnosis of pre-diabetes okay)
7. Chronic renal disease (or eGFR <50 mL/min) or renal failure (defined as receipt of renal dialysis or transplant) or nephrotic syndrome
8. History of adverse reaction or contraindications associated with metformin
9. Recent history or plan for radiocontrast
10. Self-reported dementia or severe cognitive impairment
11. Receipt of blood products within 6 months before enrollment
12. History of heart disease (New York Heart Classification greater than class II; more than non-specific ST-T wave changes on the ECG)
13. History of chronic obstructive pulmonary disease
14. Poorly controlled blood pressure (systolic BP>160, diastolic BP>90 mmHg)
15. History of an immunodeficiency
16. Use of use of investigational products, antibiotics, probiotics, or systemic immunosuppressive therapy (systemic steroids) within 1 month of study start; patients who are taking these medications chronically, with no expected discontinuation during the study period would not be considered ineligible.
17. Treatment with anticoagulants (warfarin)
18. Donated blood within the last 2 months
19. Subject is considered unsuitable for the study in the opinion of the investigator for any other reason

Ages: 63 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Change in antibody responses to PCV13 | Change from 4 weeks to 8 weeks
  The primary outcome will be antibody responses to PCV13. Antibody levels of each of the 13 different serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) will be compared between the pre-treatment values and the post treatment values.

SECONDARY OUTCOMES:
Measure of immunophenotypes | Baseline, 4 weeks and 8 weeks
  The distribution of immunophenotypes will be presented descriptively at each time point for each treatment group. To determine which immunophenotypes differed between MET and placebo groups, changes will be determined using within-patient cell count ratios for each measured phenotype between baseline and 6-weeks of study drug treatment and between baseline and the 30 days after PCV13.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lee, PhD, Principal Investigator — UT Health San Antonio
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No